CLINICAL TRIAL: NCT06336785
Title: A Prospective Clinical Trial Evaluating the "Kiss and Smile HIT" (Holistic Individualized Treatment) Algorithm
Brief Title: Kiss and Smile HIT (Holistic Individualized Treatment)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-2023-HIT-K&S
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Aesthetic
Keywords: Hyaluronic Acid; Aesthetic Injection; Holistic Individualized Treatment; Perioral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Restylane Filler Line and Dysport Neuromodulator (Experimental): This study will consist of an open-label, prospective, cohort trial design. Twenty-four subjects will be recruited.
  Subjects will be recruited based on their primary deficit, 8 subjects will have a primary deficit in lip volume, 8 subjects will have a primary deficit in lip framing and 8 subjects will have a primary deficit in expression. All subjects will receive active treatment with hyaluronic acid at Baseline, with an optional touch at week two. There will be no placebo or no-treatment control groups. Subjects will be followed for five months.
  Interventions: Device: Restylane line of soft tissue fillers and Dysport neuromodulator

INTERVENTIONS:
Device: Restylane line of soft tissue fillers and Dysport neuromodulator — Subjects will be treated with a range of hyaluronic acid-based soft tissue fillers (Restylane line) and Dysport neuromodulator

SUMMARY:
The "Holistic Individualized Treatment" (HIT) approach is used to identify treatment priorities, focus areas, and appropriate products for soft tissue filler treatments.

The "Kiss and Smile HIT" considers lip volume, lip framing and expression to improve patients appearance. This trial will assess the effectiveness of the Kiss and Smile HIT algorithm in treating patients with different kiss and smile related issues (e.g. volume loss, lips lack proper framing, lack of a confident smile due to issues with expression).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily sign and date an informed consent, including the photography addendum allowing unrestricted use of photographs for the use of marketing and educational purposes, approved by an independent ethics committee, prior to the initiation of any screening or study-specific procedures.
2. Subjects must at least 18 years old
3. Male or female
4. Subjects must be willing and able to comply with procedures required in the protocol
5. Subjects must be in good health as per investigator's judgment based on medical history
6. Female subjects of child-bearing potential must have a negative urine pregnancy test prior to any dose of study product
7. Female subjects of childbearing potential must practice at least 1 protocol-specified method of birth control that is effective from Baseline through at least 30 days after the last dose or until the end of study, whichever is longer. Female subjects of nonchildbearing potential do not need to use birth control.

Exclusion Criteria:

1. Uncontrolled systemic disease
2. Subjects do not present with or have a history of any medical condition that may place the subject at increased risk following exposure to hyaluronic acid or interfere with the study evaluation, including:

   * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
   * History of facial nerve palsy
   * Infection or dermatological condition at the treatment injection sites
   * Marked facial dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin
3. History of clinically significant medical conditions or any other reason that the investigator determines would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study medical device
4. History of an allergic reaction or significant sensitivity to constituents of the study medical device (or its excipients)
5. Subject has tattoos, jewelry, or clothing which obscure temporal region and cannot be removed
6. Subject has anticipated need for surgery or overnight hospitalization during the study.
7. History of surgical procedures in the face including any lifting procedure (e.g., facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
8. Subject has a history of facial treatment with semi- permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
9. Subjects is presenting with porphyria
10. Subjects has present with active disease, such as inflammation, infection or tumors, in or near the intended treatment sites
11. Subject has bleeding disorders or take thrombolytics or anticoagulants
12. Subjects has had known active COVID infection within 30 days of treatment
13. Female subjects that are pregnant or breastfeeding and are considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
14. Subjects has been treated with any investigational drug within 30 days prior to the first dose of study drug or is currently enrolled in another clinical study.
15. Subject must take immunosuppressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | Baseline to Week 2, Week 4, Week 8, Week 20
  Frequency of subjects having at least "improved" (e.g., "improved", "much improved" or "very much improved") on the Global Aesthetics Improvement Scale (GAIS), as graded by a blinded evaluator. Grading value varies from worse (grading of -1) to very much improved (grading of 3).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No